CLINICAL TRIAL: NCT00303602
Title: BMI Evaluation: Placebo and Active Comparator Trial of Olanzapine Zydis Pills Used Sublingually (PLATYPUS)
Brief Title: Comparing the Effect of Under the Tongue Olanzapine Versus Swallowed Olanzapine on Body Mass Index (A Ratio of Weight to Height)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10268; F1D-CA-S063
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental): Sublingual orally disintegrating olanzapine (SODO)
  Interventions: Drug: Sublingual orally disintegrating olanzapine (SODO)
- B (Active Comparator): Oral olanzapine
  Interventions: Drug: Oral olanzapine

INTERVENTIONS:
Drug: Sublingual orally disintegrating olanzapine (SODO) — 5 to 20mg dose, supplied in 5mg tablet strength, tablet should be placed under tongue for at least 60 seconds, daily for 16 weeks.
  Other Names: LY170053; Zydis
  Arms: A
Drug: Oral olanzapine — 5 to 20mg dose, supplied in 5mg tablet strength, oral administration (tablets swallowed), daily for 16 weeks.
  Other Names: LY170053; Zyprexa
  Arms: B

SUMMARY:
This study is testing if under the tongue olanzapine for schizophrenia, related psychosis, schizoaffective disorder or bipolar disorder will have less weight gain than olanzapine that is swallowed, in patients who are already gaining weight on olanzapine.

ELIGIBILITY:
Inclusion Criteria (Patients must):

* Be at least 18 years old
* Have gained weight while taking olanzapine
* Be able to visit the doctor's office seven times over 4 months (17 weeks)

Exclusion Criteria (Patients must NOT):

* Have started a weight loss program within the last 8 weeks
* Have an illness that might affect patient's weight during the study
* Have an allergy to phenylalanine, mannitol or saccharine
* Be taking any medication (except for olanzapine) that might affect patient's weight

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
- Canada (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Penticton, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dartmouth, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sydney, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chatham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greater Sudbury, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Windsor, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amersfoort
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico

REFERENCES:
- [Derived] Case M, Treuer T, Karagianis J, Hoffmann VP. The potential role of appetite in predicting weight changes during treatment with olanzapine. BMC Psychiatry. 2010 Sep 14;10:72. doi: 10.1186/1471-244X-10-72. PMID 20840778
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- SODO: Sublingual orally disintegrating olanzapine (SODO); 5 to 20 mg dose, supplied in 5 mg tablet strength, tablet should be placed under tongue for at least 60 seconds, daily for 16 weeks
- SOT: Standard oral olanzapine tablet; 5 to 20 mg dose, supplied in 5 mg tablet strength, oral administration (tablets swallowed), daily for 16 weeks
Period: Overall Study
Arm/Group | SODO | SOT
Started | 84 | 65
Completed | 65 | 50
Not Completed | 19 | 15
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 5 | 2
Not completed — Protocol entry criteria not met | 2 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Noncompliance | 2 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SODO | SOT | Total
Number analyzed (Participants) | 84 | 65 | 149
Age Continuous [Mean (Standard Deviation); unit: years] | 38.6 (13.13) | 38.7 (12.23) | 38.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 48 | 33 | 81
Region of Enrollment [Number; unit: participants]
  United States | 23 | 18 | 41
  Mexico | 27 | 23 | 50
  Canada | 29 | 21 | 50
  Netherlands | 5 | 3 | 8
Presence of Metabolic Syndrome [Number; unit: participants]
  No | 64 | 49 | 113
  Yes | 18 | 16 | 34
  Unknown | 2 | 0 | 2
Psychiatric Illness [Number; unit: participants]
  Schizophrenia | 46 | 36 | 82
  Schizophreniform | 7 | 2 | 9
  Schizoaffective disorder | 3 | 12 | 15
  Other related psychiatric disorder | 1 | 1 | 2
  Bipolar disorder | 27 | 14 | 41
Race/Ethnicity [Number; unit: participants]
  African Descent | 11 | 4 | 15
  Caucasian | 42 | 36 | 78
  East/Southeast Asian | 2 | 1 | 3
  First Nations | 2 | 0 | 2
  Hispanic | 27 | 23 | 50
  Other | 0 | 1 | 1
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic Blood Pressure | 120.3 (16.45) | 119.0 (12.49) | 119.7 (14.82)
  Diastolic Blood Pressure | 77.6 (9.62) | 75.8 (9.15) | 76.8 (9.43)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters-squared] | 28.0 (5.63) | 28.3 (4.76) | 28.1 (5.26)
Clinical Global Impression-Severity Scale [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
  units on a scale | 3.0 (0.78) | 3.2 (0.85) | 3.1 (0.81)
Fasting Glucose [Mean (Standard Deviation); unit: millimole/Liter] | 5.1 (0.77) | 5.0 (0.46) | 5.1 (0.65)
Fasting Insulin [Mean (Standard Deviation); unit: micro International Unit/milliliter] | 13.5 (14.65) | 10.0 (7.18) | 11.9 (12.06)
Fasting Lipoproteins [Mean (Standard Deviation); unit: millimole/Liter]
  Total Cholesterol | 5.1 (1.01) | 5.1 (1.01) | 5.1 (1.0)
  High-Density Lipoprotein Cholesterol | 1.2 (0.40) | 1.3 (0.34) | 1.3 (0.37)
  Low-Density Lipoprotein Cholesterol | 3.1 (0.81) | 3.0 (0.88) | 3.1 (0.84)
  Triglycerides | 1.7 (0.77) | 1.7 (0.90) | 1.7 (0.83)
Global Assessment of Functioning Scale [Mean (Standard Deviation); unit: units on a scale] — Measures physician's judgment of a patient's overall level of functioning. Ratings are based on a scale of 1 to 100, with the following classification range: 1-10 (severely impaired) to 91-100 (superior functioning).
  units on a scale | 63.4 (12.82) | 62.5 (12.39) | 63.0 (12.60)
Glycosylated Hemoglobin [Mean (Standard Deviation); unit: percent] | 5.5 (0.45) | 5.5 (0.38) | 5.5 (0.42)
Height [Mean (Standard Deviation); unit: centimeters] | 170.0 (10.18) | 168.9 (10.23) | 169.5 (10.18)
Subjective Appetite (Visual Analog Scale) [Mean (Standard Deviation); unit: units on a scale] — Participant chooses where they think their appetite lies on a 10 centimeter line between two anchors (0 - very poor appetite and 10 - very strong appetite). The possible range of scores is 0 to 100 and represents millimeters on the 10 centimeter line.
  units on a scale | 62.5 (20.85) | 65.7 (19.24) | 63.9 (20.16)
Subjective Well-Being Under Neuroleptic Treatment - Short Form [Mean (Standard Deviation); unit: units on a scale] — Measures subjective well-being for previous 7 days. 20 items covering 5 health domains (subscales) (4 items each): emotional regulation, self-control, mental functioning, social integration, and physical functioning. Individual scores range from 1 (not at all) to 6 (very much). Subscale scores range from 4 to 24. Total score ranges from 20 to 120.
  units on a scale
    Total Score | 85.5 (15.59) | 85.6 (15.00) | 85.5 (15.28)
    Social Integration Subscale | 17.0 (4.38) | 17.0 (3.97) | 17.0 (4.19)
    Physical Functioning Subscale | 17.0 (3.53) | 17.2 (3.26) | 17.1 (3.41)
    Mental Functioning Subscale | 16.7 (4.02) | 16.7 (4.20) | 16.7 (4.09)
    Self-Control Subscale | 17.0 (3.45) | 17.3 (4.15) | 17.1 (3.76)
    Emotional Regulation Subscale | 17.6 (4.07) | 17.4 (3.82) | 17.5 (3.95)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] | 96.1 (13.24) | 97.2 (12.97) | 96.6 (13.09)
Weight [Mean (Standard Deviation); unit: kilograms] | 81.1 (18.97) | 81.2 (17.05) | 81.1 (18.10)

OUTCOME MEASURES:

1. Primary Outcome: Time Course of Change From Baseline in Body Mass Index (BMI)
Description: Body mass index is an estimate of body fat based on body weight divided by height squared. Comparison of changes at various time points throughout the study. Change = Time point value minus baseline (Visit 2) value.
Time Frame: Visit 2 (Baseline) to Visit 7 (16 Weeks)
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: kilograms/square meters
Arm/Group | SODO | SOT
Number analyzed (Participants) | 82 | 63
kilograms/square meters
  Week 2 (N=82, N=63) | 0.09 (0.06) | 0.16 (0.07)
  Week 4 (N=79, N=63) | 0.25 (0.08) | 0.27 (0.09)
  Week 8 (N=75, N=58) | 0.34 (0.12) | 0.32 (0.13)
  Week 12 (N=70, N=54) | 0.47 (0.16) | 0.54 (0.18)
  Week 16 (N=67, N=51) | 0.52 (0.18) | 0.72 (0.20)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.428, Mixed Models Analysis — P-value for Week 2 Change from Baseline. There was no adjustment for multiple comparisons
Statistical Analysis 2: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.859, Mixed Models Analysis — P-value for Week 4 Change from Baseline. There was no adjustment for multiple comparisons
Statistical Analysis 3: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.885, Mixed Models Analysis — P-value for Week 8 Change from Baseline. There was no adjustment for multiple comparisons
Statistical Analysis 4: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.784, Mixed Models Analysis — P-value for Week 12 Change from Baseline. There was no adjustment for multiple comparisons
Statistical Analysis 5: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.465, Mixed Models Analysis — P-value for Week 16 Change from Baseline. There was no adjustment for multiple comparisons

2. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Body Mass Index (BMI)
Description: Body mass index is an estimate of body fat based on body weight divided by height squared. Comparison of change from baseline to endpoint. Change = Endpoint (Week 16) minus Baseline (Week 0)
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Intention to treat with last observation carried forward
Measure: Mean (Standard Deviation); unit: kilograms/square meters
Arm/Group | SODO | SOT
Number analyzed (Participants) | 82 | 63
kilograms/square meters | 0.52 (1.49) | 0.67 (1.44)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.442, ANCOVA; Least Square Mean Change Difference = -0.19, 95% CI [-0.67 to 0.30] — Change = Endpoint minus baseline

3. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Body Mass Index (BMI) for the Treatment Completers
Description: Body mass index is an estimate of body fat based on body weight divided by height squared. Comparisons of change from baseline to endpoint between participants who completed their treatment. Change = Endpoint value minus Baseline value.
Time Frame: Visit 2 (Baseline) and Visit 7 (16 Weeks)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: kilograms/square meters
Arm/Group | SODO | SOT
Number analyzed (Participants) | 60 | 47
kilograms/square meters | 0.56 (1.59) | 0.79 (1.58)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.328, ANCOVA; Least Square Mean Change Difference = -0.32, 95% CI [-0.95 to 0.32] — Change = Endpoint minus baseline

4. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Weight
Description: Weight of undressed patient (undergarments allowed), measured preferably at the same time each day.
Time Frame: Visit 2 (Baseline) and Visit 7 (16 Weeks)
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | SODO | SOT
Number analyzed (Participants) | 67 | 51
kilograms | 1.42 (0.50) | 2.08 (0.57)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.385, Mixed Models Analysis

5. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Waist Circumference
Description: Waist circumference is measured on a bare abodomen just above the hip bone.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Intention to treat with last observation carried forward
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | SODO | SOT
Number analyzed (Participants) | 76 | 58
centimeters | 1.13 (5.25) | 0.77 (5.30)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.914, ANCOVA; Least Square Mean Change Difference = 0.10, 95% CI [-1.65 to 1.84] — Change = endpoint minus baseline

6. Secondary Outcome: Number of Patients Achieving at Least 5% Loss of Body Weight in Any Post-Baseline Period
Description: Percentage loss of body weight = 100*(postbaseline weight - baseline weight)/baseline weight
Time Frame: Visit 2 (Baseline) to Visit 7 (Week 16)
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | SODO | SOT
Number analyzed (Participants) | 84 | 65
participants
  Up to Week 2 (N=82, N=63) | 0 | 0
  Up to Week 4 (N=79, N=63) | 0 | 1
  Up to Week 8 (N=75, N=58) | 2 | 2
  Up to Week 12 (N=70, N=54) | 3 | 4
  Up to Week 16 (N=67, N=51) | 4 | 6
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.325, Fisher Exact — Up to Week 16 p-value

7. Secondary Outcome: Number of Participants Discontinuing the Trial by Visit (Week)
Description: The number of participants who discontinued by visit (non-cumulative).
Time Frame: Visit 2 (Baseline) to Visit 7 (Week 16)
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | SODO | SOT
Number analyzed (Participants) | 84 | 65
participants
  Visit 3 (Week 2) Discontinuations | 3 | 1
  Visit 4 (Week 4) Discontinuations | 3 | 1
  Visit 5 (Week 8) Discontinuations | 5 | 6
  Visit 6 (Week 12) Discontinuations | 5 | 6
  Visit 7 (Week 16) Discontinuations | 3 | 1

8. Secondary Outcome: Change From Baseline to 16 Week Endpoint in Subjective Appetite Using a Visual Analog Scale
Description: Participant chooses where they think their appetite lies on a 10 centimeter line between two anchors (0 - very poor appetite and 10 - very strong appetite). The possible range of scores is 0 to 100 and represents millimeters on the 10 centimeter line.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SODO | SOT
Number analyzed (Participants) | 82 | 63
units on a scale | -8.21 (2.26) | -5.02 (2.59)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.344, Mixed Models Analysis

9. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Blood Pressure
Description: Sitting blood pressure, taken from the same arm.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Safety population with last observation carried forward
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SODO | SOT
Number analyzed (Participants) | 74 | 55
mm Hg
  Systolic Blood Pressure | 0.1 (11.62) | -0.1 (10.83)
  Diastolic Blood Pressure | 0.3 (7.55) | 0.8 (8.35)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.708, Rank-Sum Test — Systolic Blood Pressure Change to Endpoint p-value
Statistical Analysis 2: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.453, Rank-Sum Test — Diastolic Blood Pressure Change to Endpoint p-value

10. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Fasting Lipoproteins (Total Cholesterol, High-Density Lipoprotein Cholesterol [HDL-Cholesterol], Low-Density Lipoprotein Cholesterol [LDL-Cholesterol] [Calculated], and Triglycerides)
Description: Patients should be fasting a minimum of eight hours prior to lipoprotein measurements.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Safety population with last observation carried forward
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | SODO | SOT
Number analyzed (Participants) | 74 | 57
millimole/Liter
  Total Cholesterol | 0.1 (0.74) | 0.2 (0.79)
  High-Density Lipoprotein Cholesterol | -0.0 (0.24) | -0.0 (0.24)
  Low-Density Lipoprotein Cholesterol (N=73, N=57) | 0.1 (0.66) | 0.2 (0.53)
  Triglycerides | 0.1 (0.84) | 0.0 (1.01)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.187, Cochran-Mantel-Haenszel — Total Cholesterol Change to Endpoint p-value; Ranks of change from baseline were regressed on ranks of baseline value of assay. Treatments compared using residuals of this regression in CMH test
Statistical Analysis 2: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.163, Cochran-Mantel-Haenszel — High-Density Lipoprotein Cholesterol Change to Endpoint p-value; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.323, Cochran-Mantel-Haenszel — Low-Density Lipoprotein Cholesterol Change to Endpoint p-value; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.581, Cochran-Mantel-Haenszel — Triglycerides Change to Endpoint p-value; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Baseline to 16 Week Endpoint in Fasting Plasma Glucose
Description: Patients should be fasting a minimum of eight hours prior to plasma glucose measurement.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Safety population with last observation carried forward
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | SODO | SOT
Number analyzed (Participants) | 75 | 57
millimole/Liter | 0.2 (0.79) | 0.1 (0.48)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.227, Cochran-Mantel-Haenszel; [statistical method as in outcome 10, analysis 1]

12. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Fasting Serum Insulin
Description: Patients should be fasting a minimum of eight hours prior to serum insulin measurement.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Safety population with last observation carried forward
Measure: Mean (Standard Deviation); unit: microIU/milliliter
Arm/Group | SODO | SOT
Number analyzed (Participants) | 65 | 52
microIU/milliliter | 2.4 (17.72) | -0.1 (5.52)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.020, Cochran-Mantel-Haenszel; [statistical method as in outcome 10, analysis 1]

13. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in Glycosylated Hemoglobin
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Safety population with last observation carried forward
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SODO | SOT
Number analyzed (Participants) | 75 | 57
percent | 0.0 (0.24) | 0.0 (0.28)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.834, Cochran-Mantel-Haenszel; [statistical method as in outcome 10, analysis 1]

14. Secondary Outcome: Mean Changes From Baseline to 16 Week Endpoint Homeostasis Model Assessments of Insulin Sensitivity HOMA-S (Calculated)
Description: HOMA-S is an estimate of insulin sensitivity. The HOMA model is a computer model of the glucose insulin feedback system in the fasted state. The model consists of a number of non-linear empirical equations describing the functions of organs and tissues involved in glucose regulation.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Safety population with last observation carried forward.
Measure: Mean (Standard Deviation); unit: percent sensitivity
Arm/Group | SODO | SOT
Number analyzed (Participants) | 59 | 46
percent sensitivity | -18.5 (58.91) | -9.8 (62.61)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel; Ranks of change from baseline were regressed on ranks of baseline value of assay. Treatments compared using residuals on this regression in CMH test

15. Secondary Outcome: Number of Participants Meeting a Definition for the Presence of Metabolic Syndrome as Defined by Adult Treatment Panel III (ATP III) Criteria at Baseline and 16 Week Endpoint
Description: Patient meets definition of metabolic syndrome if they have >=3 risk factors: Waist circumference (men>102cm, women>88cm); triglycerides >=1.7mmol/L; HDL cholesterol (men<1.04mmol/L, women<1.30mmol/L); blood pressure >135/>=85 mmHg; Fasting glucose >=6.1mmol/L
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | SODO | SOT
Number analyzed (Participants) | 84 | 65
participants
  Baseline - Metabolic Syndrome (N=82, N=65) | 18 | 16
  Endpoint - Metabolic Syndrome (N=70, N=52) | 18 | 10
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.515, Fisher Exact — Endpoint Metabolic Syndrome p-value

16. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in the Clinical Global Impression-Severity (CGI-S) Scale
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SODO | SOT
Number analyzed (Participants) | 67 | 51
units on a scale | -0.26 (0.07) | -0.09 (0.08)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.118, Mixed Models Analysis

17. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in the Subjective Well-Being Under Neuroleptics (SWN) Scale
Description: Measures subjective well-being for previous 7 days. 20 items covering 5 health domains (subscales) (4 items each): emotional regulation, self-control, mental functioning, social integration, and physical functioning. Individual scores range from 1 (not at all) to 6 (very much). Subscale scores range from 1 to 24. Total score ranges from 1 to 120.
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SODO | SOT
Number analyzed (Participants) | 65 | 49
units on a scale | 4.79 (1.52) | 1.60 (1.73)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.161, Mixed Models Analysis

18. Secondary Outcome: Mean Change From Baseline to 16 Week Endpoint in the Global Assessment of Functioning (GAF) Scale
Description: Measures physician's judgment of a patient's overall level of functioning. Ratings are based on a scale of 1 to 100, with the following classification range: 1-10 (severely impaired) to 91-100 (superior functioning).
Time Frame: Visit 2 (Baseline) and Visit 7 (Week 16)
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SODO | SOT
Number analyzed (Participants) | 67 | 51
units on a scale | 4.61 (1.05) | 2.72 (1.20)
Statistical Analysis 1: Comparison: SODO vs SOT; Test type: Superiority or Other; p = 0.229, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | SODO | SOT
Serious Adverse Events (participants affected / at risk) | 2 | 0
Other Adverse Events (participants affected / at risk) | 32 | 32
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | SODO | SOT
Dizziness (Nervous system disorders) | 1/84 (1) | 0/65 (0)
Suicide attempt (Psychiatric disorders) | 1/84 (1) | 0/65 (0)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | SODO | SOT
Dry eye (Eye disorders) | 0/84 (0) | 1/65 (1)
Vision blurred (Eye disorders) | 0/84 (0) | 1/65 (1)
Constipation (Gastrointestinal disorders) | 3/84 (3) | 1/65 (1)
Diarrhoea (Gastrointestinal disorders) | 1/84 (1) | 0/65 (0)
Dry mouth (Gastrointestinal disorders) | 1/84 (1) | 2/65 (2)
Dyspepsia (Gastrointestinal disorders) | 1/84 (1) | 2/65 (2)
Gastritis (Gastrointestinal disorders) | 0/84 (0) | 1/65 (1)
Nausea (Gastrointestinal disorders) | 0/84 (0) | 1/65 (1)
Tongue spasm (Gastrointestinal disorders) | 0/84 (0) | 1/65 (1)
Tooth fracture (Gastrointestinal disorders) | 0/84 (0) | 1/65 (1)
Umbilical hernia (Gastrointestinal disorders) | 1/84 (1) | 0/65 (0)
Vomiting (Gastrointestinal disorders) | 1/84 (2) | 0/65 (0)
Asthenia (General disorders) | 0/84 (0) | 1/65 (1)
Fatigue (General disorders) | 3/84 (4) | 5/65 (6)
Tenderness (General disorders) | 0/84 (0) | 1/65 (1)
Eye infection (Infections and infestations) | 1/84 (1) | 0/65 (0)
Influenza (Infections and infestations) | 0/84 (0) | 2/65 (2)
Localised infection (Infections and infestations) | 0/84 (0) | 1/65 (1)
Lower respiratory tract infection (Infections and infestations) | 1/84 (1) | 0/65 (0)
Nasopharyngitis (Infections and infestations) | 1/84 (1) | 3/65 (3)
Back injury (Injury, poisoning and procedural complications) | 0/84 (0) | 1/65 (1)
Sunburn (Injury, poisoning and procedural complications) | 1/84 (1) | 0/65 (0)
Blood potassium decreased (Investigations) | 1/84 (1) | 0/65 (0)
Blood triglycerides increased (Investigations) | 1/84 (1) | 0/65 (0)
Weight increased (Investigations) | 0/84 (0) | 1/65 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3/84 (3) | 0/65 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1/84 (1) | 0/65 (0)
Increased appetite (Metabolism and nutrition disorders) | 9/84 (9) | 10/65 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/84 (0) | 2/65 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0/84 (0) | 1/65 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1/84 (1) | 0/65 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1/84 (1) | 0/65 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1/84 (1) | 0/65 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1/84 (1) | 0/65 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/84 (1) | 0/65 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1/84 (1) | 0/65 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0/84 (0) | 1/65 (1)
Akathisia (Nervous system disorders) | 2/84 (2) | 2/65 (2)
Disturbance in attention (Nervous system disorders) | 0/84 (0) | 1/65 (1)
Dizziness (Nervous system disorders) | 0/84 (0) | 4/65 (4)
Headache (Nervous system disorders) | 5/84 (6) | 5/65 (5)
Paraesthesia (Nervous system disorders) | 1/84 (1) | 1/65 (1)
Sedation (Nervous system disorders) | 0/84 (0) | 1/65 (1)
Somnolence (Nervous system disorders) | 5/84 (5) | 5/65 (6)
Syncope (Nervous system disorders) | 1/84 (1) | 0/65 (0)
Tongue paralysis (Nervous system disorders) | 1/84 (1) | 0/65 (0)
Tremor (Nervous system disorders) | 1/84 (1) | 2/65 (2)
Anxiety (Psychiatric disorders) | 3/84 (3) | 2/65 (3)
Depression (Psychiatric disorders) | 3/84 (3) | 2/65 (2)
Insomnia (Psychiatric disorders) | 2/84 (2) | 3/65 (3)
Irritability (Psychiatric disorders) | 0/84 (0) | 1/65 (1)
Libido decreased (Psychiatric disorders) | 1/84 (1) | 0/65 (0)
Psychomotor agitation (Psychiatric disorders) | 1/84 (1) | 0/65 (0)
Psychotic disorder (Psychiatric disorders) | 1/84 (1) | 0/65 (0)
Pollakiuria (Renal and urinary disorders) | 0/84 (0) | 1/65 (1)
Polyuria (Renal and urinary disorders) | 1/84 (1) | 1/65 (1)
Urinary incontinence (Renal and urinary disorders) | 0/84 (0) | 1/65 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/84 (0) | 1/65 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/84 (0) | 1/65 (1)
Rash (Skin and subcutaneous tissue disorders) | 0/84 (0) | 1/65 (1)
Haematoma (Vascular disorders) | 0/84 (0) | 1/65 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days